CLINICAL TRIAL: NCT01583504
Title: A Double Blind, Randomised Controlled Trial of High Volume Saline Injections for Chronic Midportion Achilles Tendinopathy
Brief Title: High Volume Saline Injections for Achilles Tendinopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Leeds Comunity Healthcare NHS Trust (Other)
Collaborators: National Insitute of Health Research FSF funding (Unknown)
Responsible Party: Principal Investigator, Dr Matthew Smith, Dr Matthew Smith, Leeds Comunity Healthcare NHS Trust
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11/YH/0376
Record Dates: First submitted 2012-04-20; First posted 2012-04-24 (Estimated); Last update posted 2012-04-24 (Estimated); Status verified 2012-04

CONDITIONS: Achilles Tendinopathy
Keywords: Achilles; Tendinopathy; Tendonitis; Injection
MeSH Terms: conditions — Tendinopathy | interventions — Anesthesia, Local

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- High volume saline injection (Experimental): Patients randomised to this trial arm will receive an ultrasound guided steroid and local anaesthetic injection around the achilles tendon in the same way as the control arm patients. In addition they will receive an injected bolus of normal saline (through the same needle) of between 14-25ml until the new vessels seen on ultrasound scan disappear. They will be then given a programme of stretching and strengthening exercises in the same way as patients on the control arm.
  Interventions: Procedure: Ultrasound guided injection of steroid and local anaesthetic; Procedure: High volume saline injection; Behavioral: exercise programme
- Control Arm (Active Comparator): Patients on this trial arm will receive an ultrasound guided injection of steroid and local anaesthetic between Kager's fat pad and the achilles tendon. They will then be given a programme of stretching and strengthening exercises.
  Patients on this trial arm will be offered the high volume saline injection at their 6 week follow up appointment after outcome measures have been taken by the blinded assessor. The whole cohort of patients will then be followed up at 12 and 40 weeks
  Interventions: Procedure: Ultrasound guided injection of steroid and local anaesthetic; Behavioral: exercise programme

INTERVENTIONS:
Procedure: Ultrasound guided injection of steroid and local anaesthetic — 2mls of 0.5% Bupivocaine and 25mg of hydrocortisone given as a single bolus via a 21G needle using sterile technique. The injection will be placed into the space between Kagers fat pad and the anterior aspect of the achilles tendon, into the area of maximal neovascularisation as seen on ultrasound scan.
Procedure: High volume saline injection — After steroid and local anaesthetic has been delivered, a bolus of normal saline will also be infused into the space between Kager's fat pad and the achilles tendon through the same needle, using ultrasound guidance and sterile technique. At least 14mls will be given but up to 40mls could be used. Saline will be injected until the injector determines that the appearance of neovascularisation on ultrasound has disappeared.
  Arms: High volume saline injection
Behavioral: exercise programme — a bandage will be placed on the ankle for 48 hours and instructions given to rest the ankle. The patient will be verbally shown a programme of exercises to be done over the next 6 weeks to stretch the tendon and steadily build up load bearing on it. The exercises are also clearly shown on a leaflet which the patient takes home.

SUMMARY:
Hypothesis: High volume saline injections are an effective pain relieving treatment for people with longstanding pain in the achilles tendon which has not improved with a physiotherapy programme.

Objective 1: To establish whether high volume saline injections are an effective treatment in decreasing pain for people with achilles tendinopathy

Objective 2: To investigate whether high volume saline injections can improve day to day functioning, quality of life and the ultrasound appearances of the tendon for people with achilles tendinopathy

Objective 3: To assess the tolerability of the procedure and levels of patient satisfaction using a simple questionnaire.

Objective 4: To follow up the cohort of people who have received the injection for 9 months and ascertain whether any benefits persisted, or if the symptoms recurred.

Background: Achilles tendon disorders are a common problem for athletes with a lifetime risk of around 50%. They are also common for less active people with a lifetime risk of around 6%.

Tendinopathy is a condition which is characterised by pain, difficulty with weight bearing and swelling of the tendon. Symptoms may occur with exercise at first but can progress to occurring at rest and interfering with day to day activities. When the problematic tendon is examined under the microscope, it usually shows signs of degeneration rather than inflammation - especially when symptoms have been persistent. An ultrasound scan will usually show that the tendon is swollen with an increased water content and a disorganised tendon structure.

A special type of ultrasound scan which looks at fluid flows, called a doppler ultrasound, often shows areas of increased blood flow around the tendon. Studies have shown that when these areas of increased blood flow are present, the patient tends to be experiencing more pain and stiffness in the tendon. Under the microscope, these blood vessels are often accompanied by nerve fibres and it has been suggested that these newly growing nerve endings are responsible for the persistent pain that patients experience.

There is robust evidence that a particular type of exercise programme (eccentric loading) is an effective treatment for achilles tendinopathy. These exercises involve taking weight on the tendon whilst it is being compressed rather than stretched - heel lowering exercises. Nevertheless after completing a 3 month eccentric loading exercise programme, around 24-45% of patients will still have symptoms. There is no clear consensus amongst doctors as to what is the best second line treatment to try for this group of people.

A number of different treatments have been described in research literature to try to treat this group of people with persistent symptoms, although no firm conclusion can be reached. There have been 2 small trials of high volume saline injections which showed some promising potential for the treatment. The aim of this injection is to destroy the blood vessels and nerve endings that grow into the swollen tendon to reduce pain and allow people to move and exercise more normally using the tendon. These studies simply looked at before and after injection results and did not compare the injections to a placebo or other treatment. The aim of this project is to conduct a high quality comparison of this new type of injection against a more common steroid and local anaesthetic injection around the tendon sheath. The design of the trial is a double blind, randomised controlled trial. This means that neither the patient, nor the doctor collecting data on pain scores knows which treatment the participant has been given, allowing a fair comparison of the interventions.

The main comparisons between the 2 groups will take place at a 6 week follow up appointment. Once outcome measures have been recorded by the blinded assessor, the participant will then be told which arm of the study they are on. If they previously received the control injection (steroid and local anaesthetic only)and they still have symptoms, they will at this stage be offered the high volume saline injection as well. The investigators will then follow all of the study participants up for 9 months to ascertain whether people show a persistent benefit from the treatment, or whether symptoms subsequently return.

The full study protocol is available on request from the Principle Investigator, along with information leaflets, ethical approvals etc.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+
* More than 13 weeks of pain in the achilles tendon area
* Completed eccentric tendon loading programme with a physiotherapist
* Achilles tendon tender to palpation in the midportion
* Tendon diameter greater than 0.7cm on ultrasound scan
* Evidence of neovascularisation on doppler ultrasound scan
* Sufficient English language to complete questionnaires and consent

Exclusion Criteria:

* Ultrasound evidence or previous history of partial or full tendon tear
* Another co-existing significant foot or ankle pathology
* Taking anticoagulant medication i.e: warfarin, clopidogrel, dipyridamole
* A medical condition that would affect safety of injection i.e. diabetic neuropathy, peripheral vascular disease
* Previous achilles tendon surgery
* unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2012-03; Primary Completion 2013-03 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
100mm Visual Analogue 100mm Visual Analogue Pain Score | 6 weeks post intervention
  Pain scores between the 2 trial arms are compared 6 weeks post injection

SECONDARY OUTCOMES:
Foot and Ankle Outcome Score | 6 weeks
  A validated measure of function specifically for foot and ankle conditions. Scores from the 2 trial arms are compared at 6 weeks post injection
EQ5D-3L | 6 weeks
  a widely used health status measure which will be used to compare the 2 study groups 6 weeks post injection
Diameter of symptomatic achilles tendon by ultrasound scan | 6 weeks
  the diameters of the achilles tendons will be compared at 6 weeks between the 2 trial arms
Neovascularisation grading | 6 weeks
  A grading of the amount of new vessel growth into the tendon as seen on ultrasound scan will be compared at 6 weeks between the 2 trial arms.
all outcome measures | 12 and 40 weeks
  the cohort of patients will have all outcome measures reviewed at 12 and 40 weeks to ensure resolution of symptoms

CONTACTS AND LOCATIONS:
Overall Officials: James Brown, MB ChB, Study Director — Leeds Musculoskeletal and Rehabilitation Service
Locations (1):
- Leeds Musculoskeletal and Rehabilitation Service, Leeds, W Yorks, United Kingdom